CLINICAL TRIAL: NCT03111199
Title: Influence of Cryotherapy Combined to TENS Burst in Pain, Functional Capacity and Quality of Life Patients With Non-specific Chronic Lombar Pain: A Blind Controlled Randomized Clinical Trial
Brief Title: Influence of Cryotherapy Combined to TENS Burst in Patients With Non-specific Chronic Lombar Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wouber Hérickson de Brito Vieira (Other)
Responsible Party: Sponsor-Investigator, Wouber Hérickson de Brito Vieira, Principal Investigator, Universidade Federal do Rio Grande do Norte
Organization: Universidade Federal do Rio Grande do Norte (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.953.896
Record Dates: First submitted 2017-03-17; First posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Chronic Low Back Pain
Keywords: Low back pain; Analgesia; Physical therapy
MeSH Terms: conditions — Low Back Pain; Agnosia | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Placebo Group (Placebo Comparator): The subjects of this group will be submitted to TENS bound in placebo mode in the lumbar spine.
  Interventions: Other: TENS Burst Placebo; Other: Education
- Cryotherapy Group (Experimental): The subjects of this group will be submitted to Cryotherapy in the lumbar spine.
  Interventions: Other: Cryotherpy; Other: Education
- TENS Burst Group (Experimental): The subjects of this group will be submitted to TENS Burst in the lumbar spine.
  Interventions: Other: TENS Burst Placebo; Other: Education
- TENS Burst and Cryotherapy Group (Experimental): The subjects of this group will be submitted to TENS Burst and Cryotherapy in the lumbar spine.
  Interventions: Other: Cryotherpy; Other: TENS Burst; Other: Education

INTERVENTIONS:
Other: Cryotherpy — Cryotherapy will be used by means of ice packs over a painful region. The ice will be crushed inside a bag so that it is in an ideal size that provides a coupling in a painful column in the lumbar spine; Once it has been inserted in the plastic bag and before closing it all the air must be removed to avoid a faster thawing of the ice and have difficulties of coupling.
  Arms: Cryotherapy Group; TENS Burst and Cryotherapy Group
Other: TENS Burst — The TENS Burst therapy will be performed using the KLD Sonophasys EUS 0503 electrotherapy device connected in the current therapy mode with the following parameters: 4Hz frequency, high pulse duration of 200 μsec and the current intensity will be at the maximum amplitude To generate visible muscle contraction without generating pain / discomfort. A channel will be used using self-adhesive electrodes arranged parallel to the erector muscle of the spine, so that the region to be treated is between the electrodes.
  Arms: TENS Burst and Cryotherapy Group
Other: TENS Burst Placebo — The TENS Burst placebo therapy will be performed using the KLD Sonophasys EUS 0503 electrotherapy device connected in the current therapy mode with the following parameters: 4Hz frequency, high pulse duration of 200 μsec and the current intensity will be on but without Produce the effects of visible muscle contractions because the channel will not be properly coupled in the apparatus so that the stimulation does not reach the patient. A channel will be used using self-adhesive electrodes arranged parallel to the erector muscle of the spine, so that the region to be treated is between the electrodes.
  Arms: Control Placebo Group; TENS Burst Group
Other: Education — After the electrophysical intervention, a moment of education and awareness will be held, in which the participants will receive information about the purpose of the treatment; Anatomy and biomechanics of the lumbar spine; Chronic non-specific back pain; Cognitive, emotional, genetic, social, and lifestyle factors; Intrinsic and extrinsic physical factors, biopsychosocial model: beliefs of pain and hypervigilance; Concepts of joint protection; Energy conservation and general guidelines.
  Other Names: Lesson

SUMMARY:
The purpose of this study is to analyze the effects of TENS Burst combined Cryotherapy on painful sensation, functional capacity and quality of life of patients with non-specific chronic pain.

Study hypothesis:

The TENS Burst combined with Cryotherapy offers a better response in the pain sensation, functional capacity and quality of life of patients with non-specific chronic low back pain when compared to the application of these resources in isolation.

DETAILED DESCRIPTION:
This is a blind, randomized, controlled clinical trial. The first investigator (PI) will be responsible for evaluations and reassessments; The second investigator (PII) for the process of randomization and instruction of the subjects in the intervention protocol and the third investigator (PIII) for the statistical analyzes. The study collections will take place from April 2017 until November 2017, after approval by the Ethics and Research and Qualification Committee and will be developed at the Rehabilitation Outpatient Clinic of the University Hospital Onofre Lopes - HUOL.

The investigators will select 48 individuals recruited non-probabilistically for convenience in HUOL. The sample calculation performed in G POWER software version 3.0.0.1 with 80% "power" defined the number of 40 individuals, adding to that number the 20% of possible losses during the survey. Allocation of the groups will be random, through the website http://www.randomization.com, which will include information such as sample size and number of groups. From this, the site will generate a specific coding for each group, randomly and in the form of blocks, with the following characteristics: sex, women in active cycle and use of oral contraceptives and use of analgesics. In this study, four groups will be considered: control-placebo group (gCP), cryotherapy group (gCrio), TENS Burst group (gTENSb) and Cryotherapy + TENS Burst group (gCrioTENSb). The four groups will receive educational sessions on chronic low back pain. The gCP will also undergo TENS bound in placebo mode, gCrio will undergo cryotherapy, gTENSb will undergo TENS in Burst mode and gCrioTENSb will undergo TENS Cryotherapy + Burst (combined). This protocol is in compliance with the recommendations of the Consolidated Standards of Reporting Trials - CONSORT (http://www.consort-statement.org/) for the execution of randomized clinical trials.

At the outset, all subjects will receive general instructions on the procedures to be performed, as well as information about the possible risks and benefits of all stages of the research. Individuals will then be enrolled in the survey through a specially prepared assessment form containing information on identification, sex, age, body mass index, level of education, work activity, employment status, stress, and beliefs about pain, marital status, time of onset of symptoms, presence of dermal conditions, sensitivity, ice allergy and treatment perspective. These subjects will be subject to the evaluation measures under the IP instruction, the IP will not know to which group the subjects belong. The evaluations will be performed before the 1st intervention session and will consist of the evaluation of the pain through the EVA when performing the movement and the pressure pain; Functional ability by the Roland-Morris Questionnaire, Functional Oswestry Index and Finger-to-Ground Distance; Quality of life, questionnaire SF 36 and pleasure / dissatisfaction of the intervention by Felling Scale. To maintain the blindness of the study, each individual at the time of intervention will spend 30 minutes in the intervention room and each group will have a corresponding color for the convenience of P2 (being white, blue, green and yellow).

The remaining AV2 and AV3 evaluations will be performed two days after the 10th treatment session and 4 weeks after the last treatment session, respectively, for gCP, gCrio, gTENSb and gCrioTENSb. The women will be evaluated and reassessed in the same phase, the follicular phase of the menstrual cycle to present higher thresholds of sensory perception, and will be used to identify the phases of the cycle of each volunteer following the proposed calendar method and the confirmation of regularity by, at least Less, six posterior menstrual cycles. The evaluations and interventions will be carried out in the evening shift and in the same room with a standard temperature of 24º C. A pilot study will be carried out in order to reproduce what will be done during the evaluation and intervention processes, in order to identify and correcting possible flaws with regard to the proposed procedures.

ELIGIBILITY:
Inclusion Criteria:

* Women who present a regular menstrual cycle of 21-35 days;
* Body mass index between 18.5 and 30 kg / m2;
* Low back pain for at least 12 weeks;
* Diagnosis for the treatment of chronic lumbar of non-specific origin;
* Not used electrotherapy before;
* No presenting skin alteration, vascular sensitivity or that hinder a perception of electrical stimulation and allergy to ice.

Exclusion Criteria:

* Those who are not tolerant and respect the evaluation and / or intervention procedures;
* Absence in less than two protocol treatment sessions;
* Initiate during the protocol the use of analgesics and anti-inflammatories;
* The participants to withdraw their consent to participate in the research.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-04-17 (Estimated); Primary Completion 2017-10-01 (Estimated); Study Completion 2017-11-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Pain evaluated by Visual Analog Scale at 1 month | 1 month
  Evaluated from the participants' response to pain questioning on the visual analog scale.
Change from baseline Pain evaluated by Visual Analog Scale at 2 months | 2 months
  Evaluated from the participants' response to pain questioning on the visual analog scale.
Change from baseline Pain evaluated by algometry at 1 month | 1 month
  To evaluate the pain by the pain sensation through the pressure algometer.
Change from baseline Pain evaluated by algometry at 2 months | 2 months
  To evaluate the pain by the pain sensation through the pressure algometer.study completion

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil